CLINICAL TRIAL: NCT02048930
Title: Effectiveness and Cost-effectiveness Evaluation of Easyhaler Versus Other Devices in a Real World Primary Care Population
Brief Title: Real Life Effectiveness of Easyhaler (Orion)
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: R02411
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: GPRD; effectiveness; cost-effectiveness; Easyhaler; Primary care; DPI
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Initiation cohort: Receive their first prescription for ICS therapy as one of the study drugs
  Interventions: Device: Budesonide Easyhaler; Device: Budesonide dry powder inhaler
- Step-up cohort: Receive a prescription for one of the study drugs at a dose ≥50% that of their prescribed ICS dose during baseline.
  Interventions: Device: Budesonide Easyhaler; Device: Budesonide dry powder inhaler
- Switch cohort: switch from BUD DPI (other) to BUD EH or continue on BUD DPI (other) with no change in ICS dose
  Interventions: Device: Budesonide Easyhaler; Device: Budesonide dry powder inhaler

INTERVENTIONS:
Device: Budesonide Easyhaler
Device: Budesonide dry powder inhaler

SUMMARY:
The aim of this study is to compare the clinical effectiveness and cost-effectiveness of the Easyhaler® (EH) device and other DPI devices commonly used in the UK in a UK primary care asthma population of patients aged 6 to 80 years.

DETAILED DESCRIPTION:
A recent observational study by Price et al carried out using the UK's General Practice Research Database (CPRD) to compare asthma-related outcomes for different inhaled corticosteroid (ICS) inhaler devices, using Easyhaler and dry powder inhalers (DPIs).

ELIGIBILITY:
Inclusion Criteria:

* Patients must also meet the following inclusion criteria:
* (1) Aged: 6-80 years - stratified 6-11 years; 12-60 years; ≥61 years to allow paediatrics and adolescent / adult sub analyses; and to allow for the exclusion of elderly (aged 61+) smokers and ex-smokers if required.
* (2) On-going asthma therapy: ≥2 prescriptions for asthma during the outcome period (i.e. ≥1 prescription (for any asthma therapy) in addition to the prescription for ICS at IPD (initiation / step-up/ switch).
* (3) Evidence of active asthma:

  1. Initiation - a diagnostic code for asthma
  2. Step-up / Switch - ≥2 prescriptions for asthma (at least one of which is for ICS) at different points in time during the baseline year PLUS a diagnostic code for asthma.
* (4) Have at least one year of up-to-standard (UTS) baseline data and at least one year of UTS outcome data (following the IPD).

Exclusion Criteria:

* Patients will be excluded from the analysis if they have:
* (1) Had a COPD read code at any time; and/or
* (2) Had any chronic respiratory disease, except asthma, at any time; and/or
* (3) Patients on maintenance oral steroids during baseline year; and/or
* (4) Multiple ICS prescriptions at IPD.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This will be a retrospective, observational study consisting of a one-year baseline period immediately prior to an index prescription date (IPD), and a one-year outcome period immediately following the index date.
  At the IPD, patients either:
  * Initiation cohort: receive their first prescription for ICS therapy as one of the study drugs
  * Step-up cohort: receive a prescription for one of the study drugs at a dose ≥50% that of their prescribed ICS dose during baseline.
  * Switch cohort: switch from BUD DPI (other) to BUD EH or continue on BUD DPI (other) with no change in ICS dose
Sampling Method: Non-Probability Sample
Enrollment: 24003 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
asthma control (excluding SABA usage) | 1 year
  The Composite proxy for asthma control (excluding SABA usage) during the one-year outcome period, which is defined as:
  Controlled: the absence of the following during the one-year outcome period:
  (i) Asthma-related :
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours attendance, OR
  4. Out-patient department attendance
  (ii) GP consultations for lower respiratory tract infection
  (iii) Prescriptions for acute courses of oral steroids ;
  Uncontrolled: all others.
exacerbations (ATS definition) | 1 year
  Total number of asthma exacerbations (ATS Definition) defined as an occurrence of:
  (i) Asthma-related:
  1. Hospital attendance / admissions OR
  2. A&E attendance
  (ii) Use of acute oral steroids.
exacerbations (Clinical definition) | 1 year
  Total number of asthma exacerbations (Clinical Definition) defined as an occurrence of:
  (i) Asthma-related:
  1. Hospital attendance / admissions, OR
  2. A&E attendance, OR
  (ii) GP consultations for lower respiratory related tract infections
  (iii) Use of acute oral steroids.
asthma control (including SABA usage) | 1 year
  The Composite proxy for asthma control (including SABA usage) during the one-year outcome period, which is defined as:
  Controlled: the absence of the following during the one-year outcome period:
  (iv) Asthma-related :
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours attendance, OR
  4. Out-patient department attendance
  (v) GP consultations for lower respiratory tract infection
  (vi) Prescriptions for acute courses of oral steroids ;
  Plus:
  (vii) Average prescribed daily dose ≤200mg of Salbutamol / ≤500mg of terbutaline.
  Uncontrolled: all others.

SECONDARY OUTCOMES:
treatment success definition 1 | 1 year
  Treatment Success (Definition 1) defined as:
  Successful: the absence of the following during the one-year outcome period
  (i) Asthma-related:
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours attendance, OR
  4. Out-patient department attendance
  (ii) GP consultations for lower respiratory tract infection
  (iii) Prescriptions for acute courses of oral steroids
  (iv) Any additional or change in therapy:
  1. Increased dose of ICS (≥50% increase), and/or
  2. Change in ICS and/or
  3. Change in delivery device, and/or
  4. Use of additional therapy as defined by: theophylline and leukotreine receptor antagonists (LTRAs).
  Unsuccessful: all others.
SABA dosages | 1 year
  (average daily dose during outcome year)
adherence to ICS therapy | 1 year
  categorised as: <50%, 50-<70%, 70-<100%, ≥100%.
Medication Possession Ratio (MPR) | 1 year
  The Medication Possession Ratio (MPR) for ICS is defined using the following formula.
  Medication Possession Ratio = (no. of days supply of ICS/365)x 100% The numerator is truncated at 365 if greater than 365. The MPR is a measure of adherence to therapy and a cut-off of 80% has previously been used in categorising asthma patients as adherent or non-adherent; the MPR has therefore been categorised as a dichotomous variable: < 80% and ≥ 80% for this analysis.
Treatment success (definition 2) | 1 year
  Treatment Success (Definition 2) defined as:
  Successful: the absence of the following during the one-year outcome period
  (i) Asthma-related:
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours attendance, OR
  4. Out-patient department attendance
     (ii) GP consultations for lower respiratory tract infection
     (iii) Prescriptions for acute courses of oral steroids7
     (iv) Any additional or change in therapy:
  5. Increased dose of ICS (≥50% increase), and/or
  6. Use of additional therapy as defined by: theophylline and leukotreine receptor antagonists (LTRAs).
  Unsuccessful: all others.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Principal Investigator — Research in real life